CLINICAL TRIAL: NCT00609726
Title: Prospective Evaluation of Idiopathic Pancreatitis: Role of Endoscopic Ultrasonography
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Other Study IDs: X040909004; 228552 (Other: Institutional OGCA Reference Number)
Record Dates: First submitted 2008-01-24; First posted 2008-02-07 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2015-01

CONDITIONS: Gallbladder Disease; Pancreatitis
Keywords: Endoscopic Ultrasonography; Pancreatitis; EUS
MeSH Terms: conditions — Gallbladder Diseases; Pancreatitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of the study is to determine the best evaluation for patients with idiopathic (unexplained) pancreatitis.

DETAILED DESCRIPTION:
The study evaluates the role of endoscopic ultrasonography, given that the minimally invasive procedures can diagnosis gallbladder disease as well as pancreatitis abnormalities.

ELIGIBILITY:
Inclusion Criteria:

* All patients referred to the principal investigator for unexplained pancreatitis will be enrolled.

Exclusion Criteria:

* There are no gender nor racial exclusion.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men and women diagnosed with unexplained pancreatitis.
Sampling Method: Non-Probability Sample
Enrollment: 199 (Actual)
Dates: Start 2015-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of current clinical practice for patients with idiopathic pancreatitis | 3 hours

CONTACTS AND LOCATIONS:
Overall Officials: Charles M Wilcox, M.D., Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Wilcox CM, Seay T, Kim H, Varadarajulu S. Prospective Endoscopic Ultrasound-Based Approach to the Evaluation of Idiopathic Pancreatitis: Causes, Response to Therapy, and Long-term Outcome. Am J Gastroenterol. 2016 Sep;111(9):1339-48. doi: 10.1038/ajg.2016.240. Epub 2016 Jun 21. PMID 27325219